CLINICAL TRIAL: NCT06333028
Title: A Non-interventional, Prospective, Multicenter, Single Arm, Post-Marketing Clinical Study to Evaluate the enVista® Aspire (EA) Intraocular Lens in Subjects Undergoing Cataract Extraction.
Brief Title: A Study to Evaluate the enVista® Aspire (EA) Intraocular Lens in Subjects Undergoing Cataract Extraction
Status: Completed | Type: Observational
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 938
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- enVista Aspire intraocular lens (IOL): Subjects bilaterally implanted with enVista Aspire EA IOLs.
  Interventions: Device: enVista Aspire EA IOLs

INTERVENTIONS:
Device: enVista Aspire EA IOLs — Subjects bilaterally implanted with enVista Aspire EA IOLs

SUMMARY:
A Study to Evaluate the enVista® Aspire (EA) intraocular lens in Subjects Undergoing Cataract Extraction

DETAILED DESCRIPTION:
A Non-interventional, Prospective, Multicenter, Single Arm, Post-Marketing Clinical Study to Evaluate the enVista® Aspire (EA) Intraocular Lens in Subjects Undergoing Cataract Extraction

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 22 years of age or older on the date the Informed Consent Form (ICF) is signed.
2. Subjects with a post operative BCDVA of 20/40 or better.
3. Subjects must have the capability to understand and provide written informed consent on the Institutional Review Board (IRB) approved ICF and authorization as appropriate for local privacy regulations and willing and able to comply with the follow-up study visit.
4. Subjects implanted bilaterally with enVista Aspire EA IOLs, powers ranging from + 6 to + 34.0 D, prior to enrollment into the study on or after 1 November 2023.
5. All subjects with a visually significant PCO (BCDVA worse than 20/40) who undergo a YAG capsulotomy may be enrolled 30 days post YAG procedure and with a postoperative BCDVA 20/40 or better.

Exclusion Criteria:

1. Subjects with any serious ocular pathology or underlying systemic medical disease (e.g., uncontrolled diabetes) or circumstance that, based on the Investigator's judgment, could confound the results of the study.
2. Subjects for whom a Toric IOL is indicated to achieve emmetropia.
3. Subjects for whom monovision treatment is planned.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population at study site locations
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Mean binocular BCDVA (logMAR) at Visit 1 | Day 60 to Day 270 after second eye implantation
  Mean binocular best-corrected distance visual acuity (BCDVA) (logMAR) at Visit 1. Photopic BCDVA measured at 4 meters.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - SITE 104, Dover, New Jersey
  - Site 105, Woodland Park, New Jersey
  - Site 103, Garden City, New York
  - Site 107, Cranberry Township, Pennsylvania
  - Site 106, Charleston, South Carolina
  - Site 101, Sugar Land, Texas
  - Site 102, Mount Pleasant, Wisconsin

IPD SHARING:
Plan to Share IPD: No